CLINICAL TRIAL: NCT03169010
Title: Registration Study for Rare Type of Pulmonary Hypertension
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhi-Cheng JING, MD, Director of Thrombosis and Hemostasis Center of Chinese Academy of Medical Sciences Fuwai Hospital, China National Center for Cardiovascular Diseases
Other Study IDs: RarePH135
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Hypertension
Keywords: registry; pulmonary hypertension; survival; biomarker; whole genome sequencing
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — All subjects will have a sample of blood taken for Sanger or whole genome sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Idiopathic Pulmonary Artery Hypertension: Investigators will conduct laboratory biomarker analysis and genetic analysis to identify pathogenesis or factors related to idiopathic pulmonary artery hypertension (PAH).
  Interventions: Other: laboratory biomarker analysis; Genetic: Genetic analysis
- Hereditary PAH: Investigators will conduct laboratory biomarker analysis and genetic analysis to identify pathogenesis or factors related to hereditary PAH.
  Interventions: Other: laboratory biomarker analysis; Genetic: Genetic analysis
- Hereditary Hemorrhagic Telangiectasia: Investigators will conduct laboratory biomarker analysis and genetic analysis to identify pathogenesis or factors related to hereditary hemorrhagic telangiectasia associated PAH.
  Interventions: Other: laboratory biomarker analysis; Genetic: Genetic analysis
- Pulmonary Veno-Occlusive Disease (PVOD): Investigators will conduct laboratory biomarker analysis and genetic analysis to identify pathogenesis or factors related to PVOD.
  Interventions: Other: laboratory biomarker analysis; Genetic: Genetic analysis
- Pulmonary Capillary Hemangiomatosis: Investigators will conduct laboratory biomarker analysis and genetic analysis to identify pathogenesis or factors related to pulmonary capillary hemangiomatosis associated PAH
  Interventions: Other: laboratory biomarker analysis; Genetic: Genetic analysis
- Cavernous Transformation of Portal Vein: Investigators will conduct laboratory biomarker analysis and genetic analysis to identify pathogenesis or factors related to cavernous transformation of portal vein associated PAH
  Interventions: Other: laboratory biomarker analysis; Genetic: Genetic analysis
- CTEPH: Investigators will conduct laboratory biomarker analysis and genetic analysis to identify pathogenesis or factors related to chronic thromboembolism pulmonary hypertension (CTEPH).
  Interventions: Other: laboratory biomarker analysis; Genetic: Genetic analysis
- Pulmonary Takaysu Arteritis: Investigators will conduct laboratory biomarker analysis and genetic analysis to identify pathogenesis or factors related to Pulmonary Takaysu Arteritis.
  Interventions: Other: laboratory biomarker analysis; Genetic: Genetic analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Laboratory results will be analysed to identify disease related biomarkers.
Genetic: Genetic analysis — Gene sequencing results will be analysed to identify disease related mutations.

SUMMARY:
The knowledge on the rare type of pulmonary hypertension which can not be explained by left heart disease, respiratory disease or congenital heart disease is very limited. Investigators aim to setup a national registration study for the rare type of pulmonary hypertension, to understand the natural history, survival, progression, genetic and environmental contributions to disease.

DETAILED DESCRIPTION:
The main research contents of this registration study includes:

1. Build a baseline database of the rare type of pulmonary hypertension. Collect general information, on-set symptoms and time, laboratory examination, imaging results, right heart catheterization and treatment information.
2. Follow up recruited patients at regular intervals（6m~1y). Collect information on change in patients condition, laboratory test and treatment.
3. Conduct genetic testing for gene mutation related or hereditary pulmonary hypertension. Link the clinical database to genetic database.
4. Establish bio-bank for serum/plasma, urine, stool, tissues or cells.
5. Establish prognostic study based on the clinical follow-up and genetic database.
6. Draw diagnostic and treatment algorithm for the rare type of pulmonary hypertension.

Controls subjects: blood sample and medical data collected once.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Patients diagnosed as idiopathic pulmonary artery hypertension, hereditary pulmonary artery hypertension, hereditary hemorrhagic telangiectasia associated pulmonary artery hypertension, pulmonary veno-occlusive disease, pulmonary capillary hemangiomatosis associated pulmonary artery hypertension, cavernous transformation of portal vein associated pulmonary artery hypertension, special type of congenital heart disease associated pulmonary artery hypertension, chronic thromboembolism pulmonary hypertension.
* All patients should have undergone right heart catheterization, diagnosed according to the guideline.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Patients unwilling or unable to provide written consent for participation in the study.
* Not suffering from the rare type of pulmonary artery hypertension;

Inclusion criteria-Controls

* Participant is willing and able to give informed consent for participation in the study.
* Self-reported to be healthy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Rare type of pulmonary artery hypertension
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-05-06 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival Rate of Participants | up to 10 years, at 12 months interval
Lung transplantation | up to 10 years, at 12 months interval
Change in New York Heart Association (NYHA) functional class | up to 10 years, at 3 months interval
Change in 6 mint walk distance | up to 10 years, at 3 months interval

SECONDARY OUTCOMES:
Genetic alteration in participants with rare type of PH | Baseline
  To identify the major genetic alterations in participants with rare type of PH
Change in NT-proBNP | up to 10 years, at 3 months interval
Change in hemodynamics | up to 10 years, at 6 months interval
Change in cardiac function | up to 10 years, at 3-6 months interval
  Measured by Cardiac MRI
Pulmonary endarterectomy (PEA) | up to 10 years, at 6 months interval
  e.g. operated versus non-operated
Balloon pulmonary angioplasty (BPA) | up to 10 years, at 6 months interval
  e.g. BPA versus non-BPA
Medical treatment | up to 10 years, at 6 months interval
  e.g. mono- versus combination therapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Cheng JING, MD. PhD., Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences Fuwai Hospital and Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Consent for sharing of non identifiable study data for regulatory authorities.

REFERENCES:
- [Background] Galie N, Corris PA, Frost A, Girgis RE, Granton J, Jing ZC, Klepetko W, McGoon MD, McLaughlin VV, Preston IR, Rubin LJ, Sandoval J, Seeger W, Keogh A. Updated treatment algorithm of pulmonary arterial hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D60-72. doi: 10.1016/j.jacc.2013.10.031. PMID 24355643
- [Background] Simonneau G, Robbins IM, Beghetti M, Channick RN, Delcroix M, Denton CP, Elliott CG, Gaine SP, Gladwin MT, Jing ZC, Krowka MJ, Langleben D, Nakanishi N, Souza R. Updated clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S43-S54. doi: 10.1016/j.jacc.2009.04.012. PMID 19555858